CLINICAL TRIAL: NCT06557967
Title: Prevalence of Brain Metastases and Impact on Survival in Metastatic Non-small Cell Lung Cancer by Line of Treatment
Brief Title: Study on Prevalence and Impact of Brain Metastases on Survival in Lung Cancer by Line of Treatment
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: DS1062-0003-NIS-EPI
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Non-small Cell Lung Cancer; Lung Cancer; Metastatic Cancer; Brain and Central Nervous System Cancer
Keywords: Real World Evidence; NSCLC; Brain metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasm Metastasis; Central Nervous System Neoplasms; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- mNSCLC - Overall: Participants with diagnosis of mNSCLC during study period (01/01/2015-06/30/2023)
  Interventions: Other: No drug
- mNSCLC - 1st Line of Therapy: Participants with diagnosis of mNSCLC during study period (01/01/2015-06/30/2023) treated with systemic anti-cancer therapy in first line setting.
  Interventions: Other: No drug
- mNSCLC - 2nd Line of Therapy: Participants with diagnosis of mNSCLC during study period (01/01/2015-06/30/2023) treated with systemic anti-cancer therapy in second line setting.
  Interventions: Other: No drug
- mNSCLC - 3rd Line of Therapy: Participants with diagnosis of mNSCLC during study period (01/01/2015-06/30/2023) treated with systemic anti-cancer therapy in third line setting.
  Interventions: Other: No drug

INTERVENTIONS:
Other: No drug — This is a non-interventional study and no study drug will be provided.

SUMMARY:
This study will use real-world data to assess prevalence of brain metastases in metastatic non-small cell lung cancer (mNSCLC) patients and its impact on associated clinical outcomes.

DETAILED DESCRIPTION:
This retrospective cohort database study will generate real-world evidence describing prevalence of brain metastases at metastatic diagnosis and by line of therapy, patient characteristics, treatment patterns, and clinical outcomes in metastatic non-small cell lung cancer (mNSCLC) patients

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of mNSCLC in study period (01/01/2015-06/30/2023) including newly diagnosed at metastatic stage or progression from advanced stage NSCLC
2. Age 18+ years at the time of diagnosis of mNSCLC

   Additional inclusion criteria for 1st Line of Therapy cohort:
3. Treated with systemic anti-cancer therapy in 1L setting

   Additional inclusion criteria for 2nd Line of Therapy and 3rd Line of Therapy cohorts:
4. Treated with systemic anti-cancer therapy in 2L setting treated with systemic anti-cancer therapy in 3L setting

Exclusion Criteria:

1. Evidence of other primary malignancy in the 365-day baseline period immediately prior to the first mNSCLC diagnosis in the study period
2. Evidence of stereotactic radiosurgery (SRS), stereotactic radiation therapy (SRT), or whole brain radiotherapy (WBRT) in the baseline period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with metastatic NSCLC between 2015-2023 treated with systemic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 22517 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) of (AGA+/-) mNSCLC Participant With And Without Brain Metastases by Line of Therapy | From baseline to end of follow-up or death, whichever comes first, up to approximately 40 months.

CONTACTS AND LOCATIONS:
Locations (1):
- ConcertAI Database, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No